CLINICAL TRIAL: NCT03809845
Title: Sequential High-density Surface Electromyography (HDSEMG) Recordings in Motor Neurone Disease: Fasciculations as a Biomarker of Motor Neurone Health
Brief Title: Serial Fasciculation Measurements in Motor Neurone Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KCH17-105
Record Dates: First submitted 2018-03-13; First posted 2019-01-18 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Motor Neuron Disease; Benign Fasciculation-Cramp Syndrome
MeSH Terms: conditions — Motor Neuron Disease; Neuromuscular Diseases

STUDY DESIGN:
Intervention Model Description: 20 Motor Neuron Disease (MND) patients and 5 Benign Fasciculation Syndrome (BFS) patients undergoing same assessments at 2-monthly intervals for one year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor neuron disease (Active Comparator)
  Interventions: Device: High-density surface electromyography
- Benign fasciculation syndrome (Active Comparator)
  Interventions: Device: High-density surface electromyography

INTERVENTIONS:
Device: High-density surface electromyography — High-density surface electromyography

SUMMARY:
Patients with motor neurone disease (MND) typically experience relentless motor decline and die within three years of symptom onset from respiratory muscle weakness. There are currently no effective therapies and the discovery of novel therapies is hampered by the lack of a sensitive disease biomarker. Consequently, there is a huge drive to discover novel biomarkers, which can reliably track disease progression over time. These can then be incorporated into clinical drug trials to expedite effective drug discovery.

Muscle fasciculations represent the hyperexcitability of diseased motor neurons and are almost universally present from the early stages of MND. The investigators predict that the site, frequency and shape of fasciculations might provide a sensitive measure of disease progression in an individual.

In order to calibrate this technique, the investigators will conduct a 12-month longitudinal study, recruiting 24 patients from the King's College Hospital Motor Nerve Clinic, comprising a mixture of patients with MND and those with benign fasciculation syndrome. Patients in this latter group have fasciculations but do not develop weakness and have normal lifespans. They are therefore an optimal control group. At each visit, the investigators will take resting HDSEMG recordings from all four limbs and perform standard clinical measures of disease progression. The investigators will also monitor the decline in motor unit number using a newly validated neurophysiological technique, called Motor Unit Number Index (MUNIX).

ELIGIBILITY:
Inclusion criteria for MND patients:

(i) Aged between 40 and 80 years of age inclusive, at the time of signing the informed consent.

(ii) Diagnosed with MND by a neurologist with expertise in MND.(20) For subjects with bulbar onset there must be objective limb involvement of at least one limb.

(iii) Diagnosed with MND within 24 months of symptom onset. (iv) Subjects must be ambulatory (i.e. must not be confined to a wheelchair). (v) Male and female subjects (vi) Capable of giving signed informed consent (vii) Capable and willing to comply with the requirements of the protocol (either by themselves or with assistance).

Inclusion criteria for Benign Fasciculation Syndrome (BFS) patients:

(i) Aged between 18 and 80 years of age inclusive, at the time of signing the informed consent.

(ii) Diagnosed with BFS by a neurologist with expertise in motor nerve disorders.

(iii) Male and female subjects (vi) Capable of giving signed informed consent (vii) Capable and willing to comply with the requirements of the protocol (either by themselves or with assistance).

Exclusion criteria for MND patients:

(i) Neurological (other than the subject's MND) or non-neurological co-morbidities (e.g. joint disease, respiratory disease) which limit mobility.

(ii) Clinically significant cognitive impairment in the opinion of the investigator or lacking capacity in accordance with the Mental Capacity Act (2005).

(iii) Regionally restricted forms of MND, or other atypical variants:

* Isolated corticobulbar pattern of MND with normal ambulation
* Primary lateral sclerosis
* Signs of chronic partial denervation restricted to a single limb
* MND or parkinsonism dementia complex (iv) Subjects requiring mechanical ventilation (non-invasive ventilation for sleep apnoea is allowed).

  (v) Historical or current evidence of clinically significant uncontrolled disease which, in the opinion of the chief investigator, would put the safety of the subject at risk through participation or impact the study assessments or endpoints.

(vi) Presence of an active implantable cardiac medical device (e.g., pacemaker or implantable cardioverter-defibrillator) or at a high risk for needing external defibrillation.

(vii) History of skin hypersensitivity to adhesives. (viii) Current participation in a clinical trial which in the opinion of the chief investigator might impact the objectives of this study.

Exclusion criteria for Benign Fasciculation Syndrome patients:

(i) Significant diagnostic uncertainty, whereby motor neurone disease remains a possible differential diagnosis.

(ii) Historical or current evidence of clinically significant uncontrolled disease which, in the opinion of the chief investigator, would put the safety of the subject at risk through participation or impact the study assessments or endpoints.

(iii) Presence of an active implantable cardiac medical device (e.g., pacemaker or implantable cardioverter-defibrillator) or at a high risk for needing external defibrillation.

(iv) History of skin hypersensitivity to adhesives. (v) Current participation in a clinical trial which in the opinion of the chief investigator might impact the objectives of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change in fasciculation frequency over time | 12 months
  To characterise the frequency of fasciculations in patients with motor neurone disease and to determine whether these parameters correlate with the trajectory of disease progression over a 12-month period.

SECONDARY OUTCOMES:
Change in fasciculation morphology over time | 12 months
Change in Functional Rating Scale (FRS) over time | 12 months
  Maximum score of 48; lower scores indicate worse disability
Change in motor unit number index measurements over time | 12 months
Change in MRC power sum score over time | 12 months
Change in slow vital capacity over time | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom